CLINICAL TRIAL: NCT00905502
Title: Intraoperative Fluid Management in Laparoscopic Bariatric Surgery - Does it Make a Difference?
Brief Title: Intraoperative Fluid Management in Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Idit Matot, Sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-09-IM-38590207-CTIL
Record Dates: First submitted 2009-05-17; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Morbid Obesity; Acidosis; Intra-Abdominal Abscess; Hemorrhage; Reflux; Vomiting
Keywords: Obesity; fluid management; postoperative complications; bariatric surgery; hemostasis
MeSH Terms: conditions — Obesity, Morbid; Acidosis; Abdominal Abscess; Hemorrhage; Gastroesophageal Reflux; Vomiting; Obesity; Postoperative Complications | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Restricted protocol (RG) group (Experimental): Received 4 ml/kg•hr of Lactated Ringer's solution (RL) throughout the intra-operative period.
  Interventions: Drug: Lactated Ringer's solution
- 2: Liberal protocol (LG) group (Active Comparator): Received 10 ml/kg•hr of RL solution intraoperatively.
  Interventions: Drug: Lactated Ringer's solution

INTERVENTIONS:
Drug: Lactated Ringer's solution — Patients in the RG received 4 ml/kg•hr of Lactated Ringer's solution (RL) throughout the intra-operative period
  Other Names: low fluid volume
  Arms: 1: Restricted protocol (RG) group
Drug: Lactated Ringer's solution — patients in the LG received 10 ml/kg•hr of RL solution intraoperatively
  Other Names: high fluid volume
  Arms: 2: Liberal protocol (LG) group

SUMMARY:
The objective of this study is to evaluate the effects of 'high' versus 'low' volume intraoperative fluid administration (Ringer Lactate, RL) on intra- and postoperative parameters, in obese patients undergoing laparoscopic bariatric surgery (i.e., gastric bypass), in order to establish evidence-based data for perioperative fluid management in this patient population. Based on their experience as well as several reports in the literature, the investigators hypothesized that a restrictive approach to intraoperative hydration will reduce the incidence of postoperative complications and the recovery time of gastrointestinal (GI) function, and shorten hospital stay.

DETAILED DESCRIPTION:
Obesity, a chronic disease that is increasing in prevalence in adults, adolescents, and children, is now considered to be a global epidemic. The prevalence of obesity has increased markedly in the last two decades and it is now considered to be a global epidemic. In the US 65% of all adults are overweight or obese and 30% are obese. Surgery is the only effective treatment for morbid obesity, and open Roux-en-Y gastric bypass (RYGB) has become the procedure of choice for these patients.

Several studies on perioperative fluid management have reported that 'high volume' regimens may result in overhydration having deleterious effects on cardiac and pulmonary function, recovery of GI motility, tissue oxygenation, wound healing and coagulation. Most reported randomized trials suggest that perioperative fluid management has evolved to a more restricted regimen. Specifically, restricted fluid volumes applied during bariatric procedures have been shown to reduce perioperative complications (pulmonary dysfunction, hypoxia, nausea and vomiting), thereby decrease the prevalence of morbidity and mortality associated with such procedures.

We wished to evaluate in a prospective randomized study the impact of fluid management on perioperative parameters in patients undergoing a variety of laparoscopic bariatric procedures: Roux-Y Gastric Bypass (LRYGB), Biliopancreatic Diversion with Duodenal Switch (LDS), or Sleeve Gastrectomy (LSG).

Patients were randomly allocated to one of two groups receiving either 4 ml/kg•hr or 10 ml/kg•hr of RL solution throughout the intra-operative period.

The primary endpoints of the study included: mortality rate and incidence of postoperative complications, during primary hospitalization. Readmission rate to the hospital within 30 days of surgery was another primary endpoint. The secondary endpoints included time till the patient resumed drinking and consuming soft food, length of hospital stay, differences in hematocrit, creatinine concentrations and oxygen saturation in the first and third postoperative days and with discharge, and the number of patients receiving transfusion of blood and blood products.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ( >18 years) with an American Society of Anesthesiology physical status of I-III who were presenting for laparoscopic bariatric surgery, were prospectively studied.
* Patients were considered eligible if they had a BMI > 40, or > 35 and at least one comorbid condition and were scheduled to undergo one of the following laparoscopic operations:

  * Roux-Y Gastric Bypass (LRYGB)
  * Biliopancreatic Diversion with Duodenal Switch (LDS), or
  * Sleeve Gastrectomy (LSG).

Exclusion Criteria:

* Patients aged younger than 18 years.
* Patients with renal dysfunction (creatinine > 50% upper limit of normal value).
* Congestive heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
postoperative complications: mortality and morbidity (including readmissions) | 30 postoperative days (PODs)

SECONDARY OUTCOMES:
GI recovery: time until the patient resumed drinking and consuming soft food | 3 PODs
length of hospital stay | postoperative period
differences in hematocrit, creatinine concentrations and oxygen saturation in the first and third postoperative days and with discharge | primary hospitalization
the number of patients receiving transfusion of blood and blood products | 3 PODs

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Study Chair — Tel-Aviv Sourasky Medical Center; Andrei Keidar, MD, Principal Investigator — Hadassa medical organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] McGlinch BP, Que FG, Nelson JL, Wrobleski DM, Grant JE, Collazo-Clavell ML. Perioperative care of patients undergoing bariatric surgery. Mayo Clin Proc. 2006 Oct;81(10 Suppl):S25-33. doi: 10.1016/s0025-6196(11)61178-6. PMID 17036576